CLINICAL TRIAL: NCT02366364
Title: A Randomized, Double-Blind, Placebo-Controlled Multiple Oral Ascending Dose Study of the Safety, Tolerability and Pharmacokinetics of NRX-1074 in Normal Healthy Volunteers
Brief Title: Study of Safety, Tolerability and Pharmacokinetics of NRX-1074 in Normal Healthy Volunteers
Acronym: NRX-1074
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Naurex, Inc, an affiliate of Allergan plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NRX1074-C-102
Record Dates: First submitted 2015-01-29; First posted 2015-02-19 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Major Depressive Disorder
Keywords: NRX-1074; NMDA Receptor Modulator; Major Depressive Disorder; Glycine Site Modulator
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Drug: Placebo (Placebo Comparator): Single oral administration on Day 1
  Interventions: Drug: Placebo
- Drug: NRX-1074 375 mg (Experimental): Single oral administration on Day 1
  Interventions: Drug: NRX-1074 375 mg
- Drug: NRX-1074 500 mg (Experimental): Single oral administration on Day 1
  Interventions: Drug: NRX-1074 500 mg
- Drug: NRX-1074 750 mg (Experimental): Single oral administration on Day 1
  Interventions: Drug: NRX-1074 750 mg

INTERVENTIONS:
Drug: Placebo — Single oral administration of placebo consumption on Day 1
  Arms: Drug: Placebo
Drug: NRX-1074 375 mg — Single oral administration of 375 mg consumption on Day 1
  Other Names: NRX-1074 single oral dose
  Arms: Drug: NRX-1074 375 mg
Drug: NRX-1074 500 mg — Single oral administration of 500 mg consumption on Day 1
  Other Names: NRX-1074 single oral dose
  Arms: Drug: NRX-1074 500 mg
Drug: NRX-1074 750 mg — Single oral administration of 750 mg consumption on Day 1
  Other Names: NRX-1074 single oral dose
  Arms: Drug: NRX-1074 750 mg

SUMMARY:
The purpose of this study is to assess the safety and tolerability of multiple oral (PO) ascending doses of NRX-1074 in normal healthy volunteers.

DETAILED DESCRIPTION:
NRX-1074 is a N-methyl-D-aspartate (NMDA) receptor functional partial agonist with efficacy in animal models of affective disorders including major depressive disorder. The purpose of this study is to evaluate the safety and tolerability of multiple oral (PO) ascending doses of NRX-1074 as evidenced by the incidence and severity of adverse events (AEs), changes in serum chemistry, hematology, and urinalysis, changes in physical examination findings, psychotomimetic findings and subject-reported symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects
* Aged 18 to 55 years
* For female subjects, surgically sterile or at least 2 years menopausal, or using an acceptable method of birth control. If of childbearing potential, have a documented negative blood or urine pregnancy test within 24 hours prior to dosing.
* Clinical laboratory values <2 times upper limit of normal (ULN) or deemed not clinically significant by the investigator
* Ability to understand the requirements of the study, provide written informed consent, abide by the study restrictions, and agree to return for the required assessments

Exclusion Criteria:

* Human immunodeficiency virus (HIV) infection, or hepatitis or other ongoing infectious disease.
* Current evidence of alcohol abuse (greater than 4 units of alcohol on most days; 1 unit = 1/2 pint of beer, 1 glass of wine or 1 oz. of spirits), or in the option of the investigator that subject may be alcoholic.
* Current abuse of illicit substances, using the Diagnostic and Statistical Manual (DSM) IV definition of drug abuse.
* Current smoker or use of other tobacco products.
* Currently pregnant, planning to become pregnant during the course of the study, or nursing mother.
* Type I or Type II diabetes.
* Malignancy in the last 5 years, with the exception of nonmetastatic basal cell or squamous cell carcinoma of the skin or localized carcinoma in situ of the cervix.
* Currently taking prescription or over-the-counter medications including herbal therapies, within 14 days of enrollment into the study.
* History of allergy, sensitivity, or intolerance to NMDAR ligands including ketamine, dextromethorphan, memantine, methadone, dextropropoxyphene, or ketobemidone or concomitant use of such agents.
* Received another investigational drug or device within 30 days of enrollment in this study.
* Previously participated in this study.
* Psychiatric disease including major depression, bipolar disorder, anxiety, or schizophrenia, or other medical condition that, in the opinion of the investigator, would interfere with the evaluation of the study drug safety. 13) In the option of the Investigator or the Sponsor's Study Monitor, has a history of severe renal or hepatic impairment, severe active hepatic disease, or other clinically significant medical condition that may preclude safe study participation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2015-02; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | 28 days following study drug dose
  Observed side effects and changes in laboratory values

SECONDARY OUTCOMES:
Plasma pharmacokinetics Cmax | For 24 hours after drug dose on Day 1
  Cmax after administration
Plasma pharmacokinetics - Tmax | For 24 hours after drug dose on Day 7
  Tmax after administration

CONTACTS AND LOCATIONS:
Overall Officials: Mimi Van Der Leden, MD, PhD, Principal Investigator — Chicago Research Center, Inc.
Locations (1):
- Chicago Research Center, Inc., Chicago, Illinois, United States